CLINICAL TRIAL: NCT04534153
Title: The Effect of Sodium Lauryl Sulfate on the Oral Absorption of Fexofenadine in Humans
Brief Title: Excipient Effect on Drug Absorption in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-31871
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: The Impact of Excipients on Drug Absorption
MeSH Terms: interventions — fexofenadine; Sodium Dodecyl Sulfate

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, double-blind, 3-period crossover trial. Subjects will be randomized to receive fexofenadine only under Treatment Arm 1 or fexofenadine and 3 mg SLS under Treatment Arm 2 or fexofenadine and 30 mg SLS under Treatment Arm 3.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fexofenadine without SLS (Experimental): Participants will be administered by mouth with a capsule containing 120 mg fexofenadine hydrochloride and 101 mg microcrystalline cellulose
  Interventions: Drug: Fexofenadine Hydrochloride without sodium lauryl sulfate
- Fexofenadine and 3 mg SLS (Experimental): Participants will be administered by mouth with a capsule containing 120 mg fexofenadine hydrochloride, 3 mg SLS and 101 mg microcrystalline cellulose
  Interventions: Drug: Fexofenadine Hydrochloride with sodium lauryl sulfate
- Fexofenadine and 30 mg SLS (Experimental): Participants will be administered by mouth with a capsule containing 120 mg fexofenadine hydrochloride, 30 mg SLS and 101 mg microcrystalline cellulose
  Interventions: Drug: Fexofenadine Hydrochloride with sodium lauryl sulfate

INTERVENTIONS:
Drug: Fexofenadine Hydrochloride without sodium lauryl sulfate — without sodium lauryl sulfate
  Other Names: Allegra
  Arms: Fexofenadine without SLS
Drug: Fexofenadine Hydrochloride with sodium lauryl sulfate — with sodium lauryl sulfate
  Other Names: Allegra
  Arms: Fexofenadine and 3 mg SLS; Fexofenadine and 30 mg SLS

SUMMARY:
The purpose of this study is to determine if sodium lauryl sulfate (SLS), a non-drug ingredient commonly added in drug products, affect absorption of drugs that are given together with the ingredient. Investigators want to find out if drug absorption is different in people taking the drug alone compared to people taking the drug with low and high amounts of sodium lauryl sulfate at the same time.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, 3-period crossover trial. Participants will be randomized to receive a Control capsule (fexofenadine single agent) under Treatment Arm 1 or a Test 1 capsule (fexofenadine and 3 mg SLS) under Treatment Arm 2 or Test 2 capsule (fexofenadine and 30 mg SLS) under Treatment Arm 3. Investigators will assess the effect of SLS on the absorption of fexofenadine by measuring SLS and fexofenadine concentrations in plasma and stool samples and determine the change in AUC (area under the curve), Cmax and other pharmacokinetic parameters, between Treatment Arms 2 or 3 and Treatment Arm 1.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers of all ethnic groups and races.
2. Male and females between the ages of 18-64 years old, inclusive.
3. Subjects who are willing to avoid ingestion of fruit juices and citrus bioflavonoids, such as grapefruit extract, hesperidin supplement and naringin supplement, for a period extending from one week prior to the initiation of the study until its completion.
4. Written informed consent obtained from the subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Subjects with extreme obesity (BMI > 35).
2. Subjects who are allergic to fexofenadine or SLS.
3. Subjects who have hemoglobin level lower than 12 g/dL.
4. Subjects who are pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
5. Subjects with chronic constipation.
6. Subjects consuming types of food and supplements with the potential to interfere with the study objectives as judged by the Investigator.
7. Subjects taking any drugs, especially known OATP2B1 substrates (aliskiren, atenolol, celiprolol, fexofenadine, rosuvastatin and ticlopidine, etc.) except birth control hormonal medications.
8. Subjects with a condition, disease, or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data.
9. Subjects with any disease affecting or impairing the function of the liver, kidney, or heart.
10. Subjects with gastrointestinal disease, gastrointestinal disorder, or gastrointestinal surgery.
11. Subjects with known infection with HIV, Hepatitis B or Hepatitis C (as determined by questionnaire, no laboratory diagnostics concerning these diseases will be performed within the present study). Volunteers who are cured of past Hepatitis C infection are eligible to participate with a doctor's approval letter.
12. Subjects who are smokers or have smoked in the past year and/or have smoked or ingested THC/marijuana in the past week, or who are unwilling to comply throughout the study period.
13. Alcohol use on average > 2 servings/day or > 14 servings/wk (Serving size: 12oz beer/4oz wine/2oz hard liquor) in the past week or self-reported binge drinking.
14. Subjects who are currently receiving any investigational agent or who have received any investigational agents within a period of 5 half-lives of the agent prior to the initiation of the current study.
15. Subjects who have donated whole blood within 8 weeks prior to study initiation or plan to donate blood during the study period.
16. Non-English speaking.
17. Subjects with abnormal laboratory results at Screening Visit as judged by the Investigator or study physician.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Fexofenadine | 0-48 hours
  To determine whether SLS decreases the fexofenadine area under the curve (AUC) between Fexofenadine + 3 mg SLS or Fexofenadine + 30 mg SLS and Fexofenadine only.
Maximum Plasma Concentration (Cmax) of Fexofenadine | 0-48 hours
  To determine whether SLS decreases the fexofenadine Cmax between Fexofenadine + 3 mg SLS or Fexofenadine + 30 mg SLS and Fexofenadine only.

SECONDARY OUTCOMES:
Sodium lauryl sulfate plasma concentration | 0-48 hours
  To determine plasma SLS concentration in order to understand the absorption of SLS in humans
Fexofenadine stool amount | 0-48 hours
  To determine stool amount of fexofenadine and compare between the fexofenadine only arm to the 3 mg SLS and the 30 mg SLS arm.
Sodium lauryl sulfate stool amount | 0-48 hours
  To determine stool amount of sodium lauryl sulfate and compare between the fexofenadine only arm to the 3 mg SLS and the 30 mg SLS arm.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Yang, PharmD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Ucsf Ctsi Crc, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Each participant's data will be de-identified before it is shared with others who meet specified access criteria.
Time Frame: Once after publication
Access Criteria: De-identified specimens may be shared with other researchers so they can use them for, but not limited to, genomic, epigenetic, metabolomic, proteomic and transcriptomic follow-up studies.

DOCUMENTS (1):
  • Informed Consent Form (2024-07-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT04534153/ICF_000.pdf